CLINICAL TRIAL: NCT00600028
Title: Treatment of Chronic Cough in Idiopathic Pulmonary Fibrosis With Thalidomide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Maureen R. Horton, Associate Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CG-0747; CG-0747 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Idiopathic Pulmonary Fibrosis; Cough
Keywords: idiopathic pulmonary fibrosis cough
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Thalidomide, then placebo (Experimental): Participants first received Thalidomide tablet for 12 weeks. After a washout period of two weeks, they then received placebo tablet for 12 weeks.
  Interventions: Drug: Thalidomide; Drug: Placebo
- Experimental: Placebo, then Thalidomide (Experimental): Participants first received Placebo tablet for 12 weeks. After a washout period of two weeks, they then received Thalidomide tablet for 12 weeks.
  Interventions: Drug: Thalidomide; Drug: Placebo

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 50 - 100 mg by mouth daily
Drug: Placebo — Placebo 50-100 mg by mouth per day

SUMMARY:
Idiopathic Pulmonary Fibrosis (IPF) is a rapidly progressive lung disorder that is often associated with a chronic, intractable cough. The etiology of the cough associated with IPF is unclear but it is often so severe that it adversely effects the patient's quality of life. We propose that thalidomide specifically suppresses the cough associated with idiopathic pulmonary fibrosis via its anti-inflammatory properties, by suppressing the excessive functional up-regulation of sensory fibers with in the respiratory tract of patients with IPF.

This study is a Phase III, double blinded, randomized, placebo controlled, crossover trial testing the efficacy of thalidomide in suppressing the chronic cough of IPF. The primary objective of this study is to determine the efficacy of thalidomide administered daily for 12 weeks to suppress the chronic cough in patients with idiopathic pulmonary fibrosis as measured by cough specific questionnaires, scales and improved quality of life.

DETAILED DESCRIPTION:
This study is a Phase III, double blinded, randomized, placebo controlled, crossover trial testing the efficacy of thalidomide in suppressing the chronic cough of IPF. All subjects will be randomized to either begin the study receiving the active study drug - (thalidomide) or inactive drug (placebo). Study drug will be administered in escalating dose starting at 50 mg a day increasing to 100 mg a day if cough is still present after 2 weeks. Study drug will be taken by mouth at bedtime. Patients will remain on their initial treatment for 12 weeks. After 12 weeks of treatment, the subjects will be administered the Cough Specific Quality of Life Questionnaire (CQLQ), a visual cough analogue scale, and St. Georges Respiratory Questionnaire (SGRQ). In addition, investigators will collect the subjects cough diary. After 12 weeks of treatment all subjects will enter a 2 week wash-out phase in which all drugs will be discontinued. After the 2 week wash-out phase, all subjects will again be administered the Cough Specific Quality of Life Questionnaire (CQLQ), a visual cough analogue scale, and St. Georges Respiratory Questionnaire (SGRQ). In addition, investigators will collect the subjects cough diary. All subjects will then be crossed over to the other treatment arm for an additional 12 weeks of treatment. After the second 12 weeks of treatment, the subjects will be administered the Cough Specific Quality of Life Questionnaire (CQLQ), a visual cough analogue scale, and St. Georges Respiratory Questionnaire (SGRQ). In addition, investigators will collect the subjects cough diary.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic pulmonary fibrosis for >3 months <5 years
* High resolution CT scan of chest consistent with IPF within the previous 12 months
* FVC > 40% and < 90% predicted, TLC >40% <80%, DLCo >30% <90%
* Chronic Cough - cough >8 weeks
* Age >50
* Non-child bearing potential

Exclusion Criteria:

* Pregnant or lactating women
* Women of child bearing potential
* Known etiology of lung fibrosis other than IPF
* Significant respiratory toxin exposure
* Collagen Vascular Disease
* Use of narcotic anti-cough agent in last week
* significant peripheral vascular disease or neuropathy
* history of seizures
* poorly controlled diabetes
* allergy to thalidomide

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Horton, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horton MR, Santopietro V, Mathew L, Horton KM, Polito AJ, Liu MC, Danoff SK, Lechtzin N. Thalidomide for the treatment of cough in idiopathic pulmonary fibrosis: a randomized trial. Ann Intern Med. 2012 Sep 18;157(6):398-406. doi: 10.7326/0003-4819-157-6-201209180-00003. PMID 22986377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive eligible patients were recruited by the investigators from their clinics and through self-referral between February 2008 and March 2011. 98 persons contacted our study coordinator with queries about the trial, 22 from the Johns Hopkins Interstitial Lung Disease Clinic and 76 in response to the ClinicalTrials.gov Web site.
Pre-assignment Details: One participant was excluded because of an FVC>90% predicted
Groups:
- Drug Thalidomide First, Then Placebo: Drug Thalidomide 50-100mg daily in the first intervention period and placebo daily in the second intervention period (after washout period)
- Placebo First, Then Thalidomide Drug: Placebo was administered in the first interventional period and Thalidomide 50-100mg daily in the second interventional period (after washout period).
Period: First Intervention (12 Weeks)
Arm/Group | Drug Thalidomide First, Then Placebo | Placebo First, Then Thalidomide Drug
Started | 13 (Number of participants starting the first intervention (prior to washout)) | 11 (Number of participants starting the first intervention (prior to washout))
Completed | 12 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Second Intervention (12 Weeks)
Arm/Group | Drug Thalidomide First, Then Placebo | Placebo First, Then Thalidomide Drug
Started | 12 (Number of participants starting the second intervention (after a 2-week washout)) | 10 (Number of participants starting the second intervention (after a 2-week washout))
Completed | 12 | 8
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Drug Thalidomide First, Then Placebo: Drug thalidomide 50 - 100 mg daily in the first intervention period and placebo daily in the second intervention period (after washout period)
- Placebo First, Then Thalidomide Drug: Placebo was administered in the first intervention period and Thalidomide 50 - 100 mg daily in the second intervention period(After washout period)
- Total: Total of all reporting groups
Arm/Group | Drug Thalidomide First, Then Placebo | Placebo First, Then Thalidomide Drug | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (7.11) | 65.55 (7.38) | 67.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Thalidomide in Suppressing the Chronic Cough of Idiopathic Pulmonary Fibrosis Using the Cough Quality of Life Questionnaire.
Description: The primary endpoint, suppression of cough was measured by the Cough Quality of Life Questionnaire (CQLQ) to measure the effect of interventions on cough-specific quality of life.
  CQLQ consist of 28 questions about cough and its effects using Likert-like 4-point scales, with lower scores indicating less effect of cough on health related quality of life.
  CQLQ scale ranges from 28 to 112 ( The lower the value, the higher the quality of life, 28 is considered the best).
Time Frame: 6 months
Population: All participants who received the interventions and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm Thalidomide 1st, Placebo 2nd (Intervention Thalidomide): Intervention Thalidomide : thalidomide 50 - 100 mg by mouth daily in the first intervention period
- Arm Thalidomide 1st, Placebo 2nd (Intervention Placebo): Intervention Placebo : Placebo 50-100 mg by mouth per day in the second intervention period
- Arm Placebo 1st, Thalidomide 2nd (Intervention Placebo): Intervention Placebo : Placebo 50 - 100 mg by mouth daily in the first intervention period
- Arm Placebo 1st, Thalidomide 2nd (Intervention Thalidomide): Intervention Thalidomide : thalidomide 50 - 100 mg by mouth daily in the second intervention period
Arm/Group | Arm Thalidomide 1st, Placebo 2nd (Intervention Thalidomide) | Arm Thalidomide 1st, Placebo 2nd (Intervention Placebo) | Arm Placebo 1st, Thalidomide 2nd (Intervention Placebo) | Arm Placebo 1st, Thalidomide 2nd (Intervention Thalidomide)
Number analyzed (Participants) | 12 | 12 | 10 | 8
units on a scale | 47.3 (13.7) | 55.2 (14.4) | 61.6 (11.9) | 44.5 (12.5)
Statistical Analysis 1: Comparison: Arm Thalidomide 1st, Placebo 2nd (Intervention Thalidomide) vs Arm Thalidomide 1st, Placebo 2nd (Intervention Placebo); Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 4 — The values represents three months on each intervention

2. Secondary Outcome: Efficacy of Thalidomide in Suppressing the Chronic Cough of Idiopathic Pulmonary Fibrosis Using the Visual Analog Scale of Cough and the St. George Respiratory Questionnaire.
Description: The secondary endpoint, suppression of cough was measured by the visual analog scale of cough (VAS) was significantly lower during treatment with thalidomide than placebo.
  Secondary endpoints were Cough VAS - the visual analog scale of cough evaluates the severity of cough in patients with IPF.
  Visual analog scale of cough ranges from 0 to 100 (0 is considered the best).
  St. George Respiratory Questionnaire helps to evaluate cough-specific and respiratory quality of life in patients with IPF.
  St. George Respiratory Questionnaire score ranges from 0 to 100 (0 is considered the best).
Time Frame: 6 months
Population: All participants who received the interventions and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm Placebo 1st, Thalidomide 2nd (Intervention Placebo): Intervention Placebo : Placebo 50-100 mg by mouth per day in the first intervention period
Arm/Group | Arm Thalidomide 1st, Placebo 2nd (Intervention Thalidomide) | Arm Thalidomide 1st, Placebo 2nd (Intervention Placebo) | Arm Placebo 1st, Thalidomide 2nd (Intervention Placebo) | Arm Placebo 1st, Thalidomide 2nd (Intervention Thalidomide)
Number analyzed (Participants) | 12 | 12 | 10 | 8
units on a scale
  Severity of cough (VAS Score) | 30.3 (28.5) | 65.9 (23.3) | 68 (26.8) | 17.8 (9.9)
  Quality of life (SGRQ Score) | 46.4 (19.4) | 54.7 (16.9) | 58.8 (13.3) | 40.7 (9.5)
Statistical Analysis 1: Comparison: Arm Thalidomide 1st, Placebo 2nd (Intervention Thalidomide) vs Arm Thalidomide 1st, Placebo 2nd (Intervention Placebo); Test type: Superiority or Other; p = .0001, Mixed Models Analysis; Mean Difference (Final Values) = 4 — The values represents three months on each intervention

ADVERSE EVENTS:
Groups:
- Thalidomide: Thalidomide : thalidomide 50 - 100 mg by mouth daily
- Placebo: Placebo : Placebo 50-100 mg by mouth per day
Arm/Group | Thalidomide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 8/23 | 1/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thalidomide (N=23) | Placebo (N=23)
constipation (Gastrointestinal disorders) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No